CLINICAL TRIAL: NCT06685315
Title: Research on the Syndrome Characteristics of Chronic Airway Diseases (asthma, Chronic Obstructive Pulmonary Disease) Based on Intelligent Algorithm Fusion of Phenotype Omics
Brief Title: Research on the Characteristics of Chronic Airway Diseases (asthma, COPD)
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: West China Hospital (Other); Beijing Yikang Medical Technology Co., Ltd (Unknown); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Chronic Airway Disease
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Asthma Bronchiale; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Asthma; Chronic Obstructive Pulmonary Disease; Phenomics; Intelligent algorithms; Epidemiological investigation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Collect peripheral blood, bronchoalveolar lavage fluid, urine, sputum, and feces to analyze biomarkers for different syndromes of asthma and chronic obstructive pulmonary disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Participants fill out the questionnaire — Participants fill out the questionnaire

SUMMARY:
This study will to investigate the correlation between the characteristics of the population with chronic airway diseases (asthma, chronic obstructive pulmonary disease) and syndromes, in order to reveal the disease and syndrome features of the population; Secondly, screening and identifying biomarkers for asthma and chronic obstructive pulmonary disease to provide a basis for precise prevention and treatment of the disease.

DETAILED DESCRIPTION:
Chronic airway diseases are a group of non-specific chronic airway inflammatory diseases, with a heavy disease burden and serious harm to public health. Bronchial asthma and chronic obstructive pulmonary disease are the most common and representative chronic airway diseases, with significant clinical heterogeneity and unclear disease syndrome relationships. Clarifying the characteristics of asthma and chronic obstructive pulmonary disease populations, disease features, syndrome features, and their interrelationships is an important prerequisite for achieving personalized treatment and improving efficacy. Therefore, this study adopted a stratified random sampling clinical epidemiological survey method, selecting more than 10000 asthma and chronic obstructive pulmonary disease patients nationwide, and applying an optimized respiratory disease intelligent clinical research platform to collect patient population data (age, respiratory disease history, etc.), disease information (staging, grading, typing), and syndrome information (empirical, deficiency, and mixed syndrome). Using intelligent algorithms such as high-dimensional Bayesian optimization MCC-BO, T-distribution random nearest neighbor embedding, multidimensional correlation analysis, etc. to analyze the correlation between population characteristics and diseases and syndromes; Elucidate the correlation points between different stages, grades, types, and syndromes of asthma and chronic obstructive pulmonary disease. Using phenomics and adaptive multi omics global similarity fusion method to identify their biomarkers, further revealing the disease characteristics of asthma and chronic obstructive pulmonary disease populations, and guiding the precise treatment of traditional Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for asthma or COPD.
* Age of athma range from 12 years to 80 years.Age of COPD range from 18 years to 80 years.
* The investigators agreed to participate in this clinical study by voluntarily signing an informed consent form.

Exclusion Criteria:

* Patients with respiratory diseases such as interstitial lung disease, lung malignant tumor, lung infectious diseases, pneumothorax, pleural effusion, etc., which affect the syndrome differentiation.
* Patients with combining severe cardiovascular and cerebrovascular diseases, severe liver and kidney diseases, severe hematological malignancies, etc., affecting syndrome differentiation.
* Patients with delirium, dementia, various mental illnesses.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic airway disease is a group of non-specific chronic airway inflammatory diseases, among which bronchial asthma and chronic obstructive pulmonary disease are the most common and representative. There are approximately 45.7 million asthma patients aged 20 and above in China; Nearly 100 million patients with chronic obstructive pulmonary disease are over 40 years old. Traditional Chinese and Western medicine have certain advantages in preventing and treating chronic airway diseases, but there are still key issues that restrict the improvement of therapeutic effects: the complex characteristics of chronic airway diseases, unclear disease syndrome relationships, and clear disease syndrome characteristics provide a basis for precise prevention and treatment of diseases
Sampling Method: Probability Sample
Enrollment: 10545 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Phenotype of Chronic Airway Diseases | Each registered patient is measured only once at the time of registration.
  The inflammation phenotype will be determined by measuring the different proportions of eosinophils, neutrophils and mast cells in induced sputum and peripheral blood.The inflammatory phenotypes of asthma can be divided into eosinophil asthma(eosinophil > 1.01%) ， neutrophil asthma(neutrophil > 61%)， Oligocellular asthma (eosinophil > 61%)and mixed cell asthma(eosinophil > 1.01%, neutrophil > 61%).
The Traditional Chinese Medicine Syndromes of Athma | Each registered patient is measured only once at the time of registration.
  Using the "Diagnostic Criteria for Traditional Chinese Medicine Syndromes of Bronchial Asthma (2016 Edition)" to assess the TCM syndromes of asthma.
The Traditional Chinese Medicine Syndromes of COPD | Each registered patient is measured only once at the time of registration.
  Using the "Diagnostic Criteria for Traditional Chinese Medicine Syndromes of Chronic Obstructive Pulmonary Disease (2011 Edition)" to assess the TCM syndromes of COPD.
General Demographic Data | Each registered patient is measured only once at the time of registration.
  General demographic data, including name, age（years）, sex(male / female), BMI(kg/m2), occupation, smoking history (years)and drinking history(years), will be recorded.
Asthma Control Test (ACT) | Each registered patient is measured only once at the time of registration.
  ACT includes five questions. Every question will be assessed using a 5-point scale with scores ranging from 5 to 25. The higher the score, the better the symptom control.25 is considered complete control level, 20 ~ 24 is considered good control level, and <20 is considered non-control level.
COPD Assessment Test (CAT) | Each registered patient is measured only once at the time of registration.
  0-40 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was >10, the participant needed to be seen by a physician for further testing to determine if they had COPD.
Clinical Symptoms and Signs Questionnaire | Each registered patient is measured only once at the time of registration.
  Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, expectoration, chest tightness, shortness of breath, wheezing and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
modified Medical Research Council (mMRC) | Each registered patient is measured only once at the time of registration.
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
Forced Expiratory Volume in One Second (FEV1) | Each registered patient is measured only once at the time of registration.
  FEV1 will be applied to assess pulmonary function.
Forced Vital Capacity (FVC) | Each registered patient is measured only once at the time of registration.
  FVC will be applied to assess pulmonary function
Diffusing capacity of the lungs for carbon monoxide (DLCO) | Each registered patient is measured only once at the time of registration.
  DLCO will be applied to assess pulmonary function.
Cough and Sputum Assessment Questionnaire （CASA-Q） | Each registered patient is measured only once at the time of registration.
  Using the CASA-Q to assess the impact of cough and sputum on the quality of life of patients with chronic airway diseases.The questionnaire covers four domains: cough symptoms (3 items), impact of cough (8 items), sputum symptoms (3 items), and impact of sputum (6 items). Each item is scored based on frequency from "never" to "always" and intensity from "not at all" to "a lot/extremely". For each domain, the items are aggregated and rescaled to obtain a score from 0 to 100, with higher scores indicating less respiratory impairment.
Sputum Characteristic Score | Each registered patient is measured only once at the time of registration.
  Using sputum characteristics scoring to assess the impact of airway mucus hypersecretion in patients with chronic airway diseases, which mainly includes the amount of sputum, the color of sputum, the viscosity of sputum, odor, composition of sputum, and the degree of sputum expectoration.
  A comprehensive scoring scale from 1 to 5 is used, where 1 indicates normal sputum characteristics, and 5 indicates severely abnormal sputum characteristics.
Sputum Viscosity Grading | Each registered patient is measured only once at the time of registration.
  Using sputum viscosity grading to assess airway mucus hypersecretion in chronic airway diseases. Grade 0 - No sputum, Grade 1 - Thin sputum, Grade 2 - Moderately viscous sputum, Grade 3 - Highly viscous sputum.
mucin 5B（MUC5B） | Each registered patient is measured only once at the time of registration.
  Using ELISA technology to detect MUC5B in induced sputum.
mucin 5AC（MUC5AC） | Each registered patient is measured only once at the time of registration.
  Using ELISA technology to detect MUC5AC in induced sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Suyu Li Professor, Study Chair — First Affiliated Hospital of Henan University of Traditional Chinese Medicine